CLINICAL TRIAL: NCT06004609
Title: Using Large-area Low-level Light Therapy for Treating Adhesive Capsulitis of the Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202209047DIPA
Record Dates: First submitted 2023-07-16; First posted 2023-08-22 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-11

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: adhesive capsulitis; low-level laser therapy
MeSH Terms: conditions — Bursitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (low-level laser therapy with conventional physical therapy) (Experimental): Low-level laser therapy two to three times a week, 10 minutes each time, totally 24 times, for 8 to 10 weeks. Along with conventional physical therapy, two to three times a week, for 12 to 14 weeks.
  Interventions: Device: Low-level laser therapy (LLLT); Other: Conventional physical therapy
- Conventional group (conventional physical therapy only) (Active Comparator): Conventional physical therapy, two to three times a week, for 12 to 14 weeks.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Low-level laser therapy (LLLT) — Low-level laser therapy (LLLT), three time each week, 10 minutes each time, during the first 8 weeks of the treatment trial.
  Arms: Treatment group (low-level laser therapy with conventional physical therapy)
Other: Conventional physical therapy — Conventional physical therapy will be applied three time each week, for 12 weeks

SUMMARY:
Adhesive capsulitis, is a common problem characterized by the insidious onset of glenohumeral pain and limitation of shoulder motion in all planes. Clinically, frozen shoulder could be divided into freezing, frozen and thawing stage. The treatments of frozen shoulder are mainly conservative, including non-steroidal anti-inflammatory medications and physiotherapy. Due to debilitating pain at a certain stage and protracted clinical course, intra-articular corticosteroid injection in the early stages of idiopathic adhesive capsulitis has long been used to treat adhesive capsulitis with satisfactory result. However, intra-articular steroid injection still raise some controversy and is still considered too invasive for some patients.

Low-level laser therapy (LLLT) is a safe and non-invasive alternative. LLLT can employ photo-biomodulation effects to help normalize cellular functions and is considered to have partial effect in many shoulder soft tissue disorders. Possible mechanisms include increasing adenosine triphosphate production, fibroblast activity and collagen synthesis. One prospective cohort study has shown that LLLT can be effective in the management of the early phase (less than 6 weeks of disease onset) of adhesive capsulitis of the shoulder in elderly who failed to respond to conventional physical therapy and nonsteroidal anti-inflammatory medications and improvement was found maintained up to 2 years.

To this date, no randomized controlled study has been made to establish the possible role of LLLT as an adjuvant therapy on adhesive capsulitis. Also, no study has researched the effect of LLLT on patient with later stage/chronic phase of adhesive capsulitis. The objective of this paper is to report the clinical result of a study on the efficacy of LLLT as an add-on therapy in the management of adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 to 85 years old
* Diagnosed with adhesive capsulitis clinically. Painful restriction of both active and passive flexion less than 120° and 50% restriction of the external rotation aside the body
* Visual analog scale of shoulder motion pain greater than 3 on a scale of 10
* No fracture, dislocation, or arthritis in shoulder region

Exclusion Criteria:

* History of or scheduled shoulder or chest surgery
* Significant shoulder trauma within the previous 2 years
* Presence of cervical radiculopathy or other central or peripheral neurologic deficits of the upper limb
* Known shoulder tendon tear or active tendinitis or bursitis as confirmed with US
* Contraindication of low-level light therapy

  1. Pregnancy, cancer, patient with pacemaker, high bleeding tendency, or longterm corticosteroid use.
  2. Poor consciousness state, or patients with sensory impairment
  3. Patients hypersensitive to light
  4. Severe circulatory system disorder

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder range of motion | 24 weeks after enrollment
  Shoulder flexion, abduction, external rotation, internal rotation
Shoulder pain score | 24 weeks after enrollment
  Visual analogue scale for pain during shoulder motion (scale from 0 to 10, with higher scores mean worse outcome)

SECONDARY OUTCOMES:
Functional evaluation | Immediate upon enrollment, and 8, 12, 24 weeks after enrollment
  Shoulder Pain Disability Index (SPADI)
Ultrasound examination | Immediate upon enrollment, and 8, 12, 24 weeks after enrollment
  Thickness of coracohumeral ligament and inferior glenohumeral capsule
Functional evaluation | Immediate upon enrollment, and 8, 12, 24 weeks after enrollment
  Disability of the Arm, Shoulder, and Hand (DASH) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No